CLINICAL TRIAL: NCT03428191
Title: The Research About the Target Effect-site Concentration of Remifentanil Inhibiting Stress Reaction of the Perineal Prostate Puncture When Dexmedetomidine Being Continuous Pumping
Brief Title: Target Effect-site Concentration of Remifentanil in Transperineal Prostate Puncture
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese Medical Association (Network)
Responsible Party: Sponsor
Other Study IDs: MAC-0109
Record Dates: First submitted 2018-01-25; First posted 2018-02-09 (Actual); Last update posted 2018-02-09 (Actual); Status verified 2017-02

CONDITIONS: Anesthesia, Intravenous
Keywords: dexmedetomidine; remifentanil; prostate puncture and biopsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months

INTERVENTIONS:
Drug: Remifentanyl+Dexmedetomidine — In all patients, dexmedetomidine was injected at a bolus of 0.6 mg/kg and then continuously infused at 0.6 ug/kg/h using the conventional continuous microinfusion pump. the target Effect-site concentration of remifentanil was determined by sequential method.
  Other Names: target effect-site concentration of remifentanil

SUMMARY:
The research about the target effect-site concentration of remifentanil, inhibiting stress reaction of the perineal prostate puncture when Dexmedetomidine being continuous pumping

DETAILED DESCRIPTION:
Patients who were scheduled to undergo transperineal prostate puncture and biopsy were recruited into our study. In all patients, dexmedetomidine was injected at a bolus of 0.6 mg/kg and then continuously infused at 0.6 ug/kg/h using the conventional continuous microinfusion pump. the target Effect-site concentration of remifentanil was determined by sequential method. The first target effect-site concentration of remifentanil was set to 4.5ng/ml, the difference of adjacent target concentration was 0.5 ng/ml. Cardiovascular positive reaction was defined as the changes of heart rate or systolic blood pressure was more than 15% compared with baseline values, or body movement observed. The adjacent target concentration difference was adjusted to 0.2 ng/ml after 3 negative and positive reaction cycles. If the first had a cardiovascular positive reaction, the target concentration of remifentanil increased by a concentration gradient. Conversely, the target concentration of remifentanil decreased by a concentration gradient.

ELIGIBILITY:
Inclusion Criteria:

* patients of perineal prostate puncture

Exclusion Criteria:

* sinus bradycardia or atrioventricular block serious heart, brain, lung, liver, kidney, and metabolic disease allergy for dexmedetomidine or opioid

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients of perineal prostate puncture
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-02 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
the target effect-site concentration of remifentanil | intraoperative
  the target Effect-site concentration of remifentanil was determined by sequential method.

CONTACTS AND LOCATIONS:
Overall Officials: Liu Yi, D.M, Study Director — Department of Anesthesiology, Changhai Hospital Shanghai, Shanghai, China, 200433
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China